CLINICAL TRIAL: NCT05737563
Title: A Phase III, Randomized, Multicenter Study of PD-1 Antibody Combined With mXELIRI Versus mXELIRI in the Second-line Treatment of Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: PD-1 Antibody Combined With mXELIRI Versus mXELIRI in the Second-line Setting for ESCC
Acronym: Escape
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other); Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mXELIRI in ESCC
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma Abdominal Stage 0
Keywords: PD-1 inhibitor; Capecitabine; Irinotecan; Second-line; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Immune Checkpoint Inhibitors; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PD-1 Antibody Combined With mXELIRI
  Interventions: Drug: PD-1 Inhibitors; Drug: Irinotecan; Drug: Capecitabine tablets
- Control (Active Comparator): mXELIRI
  Interventions: Drug: Irinotecan; Drug: Capecitabine tablets

INTERVENTIONS:
Drug: PD-1 Inhibitors — Teripulimab 240mg, injection or Carrelizumab 200mg, injection, every 3 weeks.
  Arms: Experimental
Drug: Irinotecan — Irinotecan: 200mg/m2, injection (For patients who are confirmed to be homozygous for UGT1A1*6 or UGT1A1*28 or UGT1A1*6 and UGT1A1*28 at the same time, the starting dose of CPT-11 is 150 mg/m2).
Drug: Capecitabine tablets — Capecitabine: 1600 mg/m2/d, oral, 2 weeks on and 1 week off.

SUMMARY:
This trial is a prospective, multicenter, randomized controlled trial. The sample size was 380. Patients with advanced or metastatic esophageal squamous cell carcinoma will be randomized to receive PD1 antibody combined with mXELIRI or mXELIRI regimens in a 1:1 ratio. The stratification factors include PS status (0 vs 1), PFS of first-line treatment (PFS < 3 months versus PFS ≥3 months) . Six cycles of chemotherapy are planned every 3 weeks, for a total of 18 weeks, after which the investigator can decide whether to provide capecitabine with or without PD1 antibody maintenance therapy. Efficacy assessments were performed every 6 weeks before disease progression during treatment. Survival status was followed every 3 months after disease progression.

DETAILED DESCRIPTION:
Esophageal cancer is the seventh most common cancer and the sixth most common cause of cancer related death worldwide. Globally, there were 604,000 new cases of esophageal cancer and 544,000 deaths in 2020. China is in the high incidence area of esophageal cancer, with 253,000 new cases of esophageal cancer and 194,000 deaths in 2016. Esophageal cancer has become a malignant disease that seriously endangers the health and social development.

Squamous cell carcinoma and adenocarcinoma are common pathological types of esophageal cancer. The main risk factors for esophageal squamous cell carcinoma are smoking and alcohol consumption. Esophageal squamous cell carcinoma is the most important pathological type of esophageal cancer in China, accounting for more than 90% of esophageal cancer.

The prognosis of esophageal cancer is very poor, most patients are in the middle and advanced stages at the time of diagnosis. The natural course of the disease is only 6-8 months, and the 5-year survival rate is less than 20%. In addition, 90% of patients undergoing surgery may have recurrent metastasis, and even those with very early staging (T1) still have the risk of relapse or metastasis within 5 years. Therefore, in recent years, scholars from various countries have continued to explore effective treatment methods in order to improve the quality of life and prolong the survival of esophageal cancer patients.

Palliative chemotherapy is the mainstay of treatment for advanced metastatic esophageal cancer including paclitaxel, platinum, fluorouracil, or irinotecan. Multiple phase III clinical studies have shown that PD-1 antibodies in addition to PF (fluorouracil plus cisplatin) or TP (paclitaxel plus cisplatin) regimens can improve the effective rate and prolong PFS and OS. Therefore, PD-1 antibody combined with chemotherapy has become the new standard first-line treatment for patients with advanced esophageal cancer.

Prior to the advent of PD-1 antibodies, the second-line regimen for advanced esophageal cancer was to select drugs that were not used in first-line chemotherapy, such as taxans or irinotecans. Keynote181, Attraction-03, and ESCORT studies have suggested that PD-1 antibody monotherapy is superior to standard chemotherapy in the second-line treatment of advanced esophageal cancer. In ESCORT studies, PD-1 antibodies and conventional chemotherapy (docetaxel or irinotecan) were 20.2 percent and 6.4 percent effective, median PFS at 1.9 months, and median OS at 8.3 months and 6.2 months, respectively. Based on the above research results, China's Food and Drug Administration has approved PD-1 antibody for the second-line treatment of advanced esophageal cancer.

Therefore, we intend to design a prospective, multicenter, randomized controlled clinical study based on the characteristics of esophageal cancer in China, explore the efficacy and safety of PD-1 antibody combined with mXELIRI compared with mXELIRI in the second-line treatment of metastatic esophageal squamous cell carcinoma. We will further analyze the significance of cross-line use of PD-1 antibody and analyze the possible benefit population.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form
2. Age≥ 18 years old, gender is not limited
3. Estimated survival time≥ 3 months
4. Physical status ECOG status score of 0 or 1
5. metastatic esophageal squamous cell carcinoma, including patients with postoperative recurrence and metastasis that cannot be operated or are not suitable for radical radiotherapy, first-line chemotherapy combined with PD-1 antibody therapy is unsuccessful or intolerable (first-line chemotherapy does not use fluorouracils and irinotecan)
6. If metastatic esophageal cancer has serious clinical symptoms due to lesions, palliative radiotherapy is required first, and radiotherapy is required to be completed for more than 4 weeks (radiotherapy lesions include but are not limited to primary lesions, bones, and lymph nodes)
7. Bone marrow hematopoietic function: hemoglobin ≥ 9.0g/dL, white blood cell ≥ 4.0×109/L, neutrophil ≥ 1.5×109/L, platelet ≥ 90×109/L
8. Liver and kidney function: total bilirubin ≤ 1.5 × ULN, creatinine ≤ 1.0 × ULN, AST/ALT ≤ 2.5 ULN, ALP 5.0 ULN, creatinine clearance ≥ 60mL/min, subjects with liver metastases: AST/ALT ≤5.0 ULN
9. Female subject must have taken reliable contraceptive measures of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. and be willing to use an appropriate method of contraception during the trial and 8 weeks after the last administration of the test drug. Male subject should agree to use appropriate contraceptive methods or to have been surgically sterilized during the trial and 8 weeks after the last administration of the test drug
10. Those who have good compliance and can follow up according to the requirements of the plan.

Exclusion Criteria:

1. previous useing of fluorouracil or irinotecan for metastatic disease;
2. received radiotherapy within 4 weeks prior to enrollment;
3. patients with symptomatic brain metastases;
4. uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage (once a month or more frequently); Multi-segment vertebral bone metastasis, easy to cause fracture, risk of paraplegia bone metastasis patients. Except for patients who are assessed by a specialist to be stable and do not need to be treated for the time being;
5. Patients who are known to have complete endoscopic obstruction and require interventional treatment or surgery to relieve obstruction and who have undergone tracheal or esophageal stenting;
6. Can not take oral medication;
7. BMI less than 17.5kg/m2, weight loss of >10% within about 2 months before the first administration of study treatment (need to consider a large number of pleural ascites changes) or other indicators show severe malnutrition;
8. Those who are allergic to the drugs used in this program or their components;
9. patients receiving chronic or multi-dose corticosteroid therapy (inhaled steroids or short-term oral cortisol as clinically indicated are allowed);
10. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-related vascular thrombosis, Wegener's granulomatous disease, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, glomerulonephritis, etc. Patients who are hypothyroid but receiving a stable dose of thyroid hormone replacement therapy may be enrolled in this study; Patients with type 1 diabetes who are treated with a stable dose of insulin dosing regimen and whose blood glucose is controlled may be enrolled in this study;
11. Patients with positive human immunodeficiency virus (HIV) test results
12. Patients with active pulmonary tuberculosis (clinical diagnosis includes clinical history, physical examination and imaging findings, and TB examination according to local medical practice);
13. received oral or intravenous antibiotics within 2 weeks prior to randomization; Patients receiving prophylactic antibiotic therapy (eg, to prevent urinary tract infection or to prevent exacerbation of chronic obstructive pulmonary disease) may be enrolled.
14. Important cardiovascular diseases, such as heart disease (grade II or higher) as defined by the New York College of Cardiology, myocardial infarction within 3 months prior to randomization, unstable arrhythmia, unstable angina, cerebrovascular accident or transient ischemic attack; 50% of patients with known coronary artery disease, congestive heart failure that does not meet the above criteria, or left ventricular ejection fraction < must be treated with a stable regimen deemed best by the attending physician, and if necessary, a cardiologist;
15. Chronic hepatitis B carriers with untreated chronic hepatitis B or HBV DNA > 1000 IU/mL at the time of screening. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 1000 IU/mL) can be enrolled;
16. Had major surgery (other than diagnostic surgery) within 28 days prior to randomization, or was expected to undergo major surgery during the study period;
17. Previous allogeneic bone marrow transplantation or solid organ transplantation;
18. Patients with serious complications, such as active gastrointestinal bleeding, perforation, jaundice, gastrointestinal obstruction, and active infection; Including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc.; history of idiopathic pulmonary fibrosis, organising pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, interstitial pneumonia, or evidence of active pneumonia on chest CT scan screening;
19. Neurological or psychiatric abnormalities affecting cognitive ability;
20. pregnant or lactating women;
21. Those who have participated in other clinical studies in the past 30 days;
22. Previous PD1 antibody therapy with grade 3 immune-related adverse reactions greater than or equal to 3
23. Patients with other primary malignant tumors other than esophageal cancer (except cured skin basal cell carcinoma and cervical carcinoma in situ);
24. Any other disease, metabolic disorder, abnormal result of physical examination or laboratory test that has reason to suspect may lead to contraindications to the use of the investigational drug, or affect the reliability of the results of the study, or put the patient at high risk of treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 1 year
  The time from registration to death due to any cause, or censored at date last known alive.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 1 year
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Objective response rate (ORR) | Up to 6 months
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
Disease Control Rate (DCR) | Up to 6 months
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, GD, China

IPD SHARING:
Plan to Share IPD: No